CLINICAL TRIAL: NCT03730727
Title: Maximizing Postprandial Glycaemic Control: When is the Right Time for Physical Activity
Brief Title: Exercise-meal Timing and Postprandial Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ERN_18-0942
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia, Postprandial; Physical Activity; Glucose Intolerance
Keywords: Exercise; Type 2 diabetes; Walking; Standing; Circuit exercises; Inactivity; Blood glucose control; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Motor Activity; Glucose Intolerance; Sedentary Behavior | interventions — Exercise; Meals

STUDY DESIGN:
Intervention Model Description: Three independent groups of participants will enter 1 of 3 studies, each of which involves a randomised, crossover, controlled trial containing 4 trials: (i) control, meal ingestion no activity; (ii) activity bout immediately prior to meal; (iii) activity bout immediately after ingestion of meal; (iv) activity bout 30-mins after ingestion of meal.
Who Masked: Outcomes Assessor
Masking Description: Although the trial order will be randomized, it is not possible to blind the participant or the investigator to the timing between meals and physical activity. However, the trial allocation and order will be blinded to the outcomes assessor when statistical analyses are performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): A liquid meal replacement shake containing 500 kcal (55% kcals from carb, 30% fat, 15% protein) will be administered at approx. 8 am following an 8-10 hour overnight fast. Postprandial blood glucose responses will be assessed for 2-hours post-ingestion. Two-hours after ingestion of the meal, participants will complete a bout of physical activity (either 30-mins of standing still, 30-mins of walking at a self-selected brisk pace on a treadmill, or 3-sets of circuit-exercises [10 squats, 10 push-ups, 10 lunges, 10 sit-ups]).
  Interventions: Behavioral: Physical activity; Dietary Supplement: Meal
- Immediate prior to meal (Experimental): At approx. 8 am following an 8-10 hour overnight fast, participants will complete a bout of physical activity (either 30-mins of standing still, 30-mins of walking at a self-selected brisk pace on a treadmill, or 3-sets of circuit-exercises [10 squats, 10 push-ups, 10 lunges, 10 sit-ups]). Immediately after completion of this bout, a liquid meal replacement shake containing 500 kcal will be administered. Postprandial blood glucose responses will be assessed for 2-hours post-ingestion.
  Interventions: Behavioral: Physical activity; Dietary Supplement: Meal
- Immediate post-meal (Experimental): A liquid meal replacement shake containing 500 kcal will be administered at approx. 8 am following an 8-10 hour overnight fast. Postprandial blood glucose responses will be assessed for 2-hours post-ingestion. Immediately after ingestion of the meal, participants will complete a bout of physical activity (either 30-mins of standing still, 30-mins of walking at a self-selected brisk pace on a treadmill, or 3-sets of circuit-exercises [10 squats, 10 push-ups, 10 lunges, 10 sit-ups]).
  Interventions: Behavioral: Physical activity; Dietary Supplement: Meal
- 30-minutes post-meal (Experimental): A liquid meal replacement shake containing 500 kcal will be administered at approx. 8 am following an 8-10 hour overnight fast. Postprandial blood glucose responses will be assessed for 2-hours post-ingestion. Thirty-minutes after ingestion of the meal, participants will complete a bout of physical activity (either 30-mins of standing still, 30-mins of walking at a self selected brisk pace on a treadmill, or 3-sets of circuit-exercises [10 squats, 10 push-ups, 10 lunges, 10 sit-ups]).
  Interventions: Behavioral: Physical activity; Dietary Supplement: Meal

INTERVENTIONS:
Behavioral: Physical activity — Physical activity will consist of either 30-mins of standing still, 30-mins of walking at a self-selected brisk pace on a treadmill, or 3-sets of circuit-exercises (10 squats, 10 push-ups, 10 lunges, 10 sit-ups).
Dietary Supplement: Meal — Liquid meal replacement shake containing 500 kcal, with 55% kcals from carb, 30% from fat, and 15% from protein.

SUMMARY:
Physical activity helps maintain optimal postprandial blood glucose control. However, there is a lack of clear information regarding the optimal meal-activity timing required to maximize blood glucose control. By using continuous glucose monitoring (CGM), this randomized controlled trial will determine whether implementing a bout of physical activity immediately before, or immediately after, or shortly after a meal is most optimal. This study will also independently examine the effects of three different physical activities: walking, standing, and circuit-exercises. Minimizing the changes in blood glucose following a meal not only reduces the risk of type 2 diabetes but also reduces cardiovascular-related mortality. Therefore, the data produced by this project will have very important implications for informing healthcare policy and physical activity recommendations.

DETAILED DESCRIPTION:
Healthy volunteers will undergo an informed consent and screening visit to determine their eligibility. Participants who are included will then be assigned to one of the three studies (walking, standing, or circuit-exercises) and then come to the lab on 5 consecutive mornings to undergo a pre-trial visit and 4 experimental trial visits (A, B, C, and D). The order of the experimental trial visits will be randomized in a counter-balanced, cross-over design.

Screening visit: Having read the participant info sheet, a study investigator will discuss the project with the potential participant who will have the chance to ask any questions. Informed consent will be sought and a General Health and Physical Activity Questionnaire will be completed. Body weight, height, resting heart rate, blood pressure, and waist circumference will be measured, and blood measures of glycated hemoglobin, triglycerides, and cholesterol will be taken.

Pre-trials visit: Participants will come to the laboratory to receive an accelerometer physical activity monitor, a continuous glucose monitor, and to complete a physical activity bout (walking, standing, or stair climbing, depending on which study they are enrolled). Over the next 5 consecutive days, participants will be instructed to maintain their normal diet and activity habits, to record their dietary intake, to refrain from vigorous exercise and alcohol, and continue wearing the accelerometer and continuous glucose monitoring devices at all times.

Experimental trial A: Following an 8-10 hour overnight fast, participants will come to the lab and will be given a 500 calorie meal-replacement drink to consume within 10 minutes. They will remain in a seated position for 2 hours and then complete the physical activity bout (30-min walk, 30-min stand, or 10-min circuit-exercises) after which they may leave the lab. Resting and post-activity heart rate and blood pressure will be recorded.

Experimental trial B: Following an 8-10 hour overnight fast, participants will come to the lab and complete the physical activity bout. Immediately after this they will be given a 500 calorie meal-replacement drink to consume within 10 minutes and will remain in a seated position for 2 hours, after which they may leave the lab. Resting and post-activity heart rate and blood pressure will be recorded.

Experimental trial C: Following an 8-10 hour overnight fast, participants will come to the lab and will be given a 500 calorie meal-replacement drink to consume within 10 minutes. Immediately after finishing the meal they will complete the physical activity bout and then remain in a seated position until 2-hours has passed since ingesting the meal. After this time they may leave the lab. Resting and post-activity heart rate and blood pressure will be recorded.

Experimental trial D: Following an 8-10 hour overnight fast, participants will come to the lab and will be given a 500 calorie meal-replacement drink to consume within 10 minutes. Thirty minutes after finishing the meal they will complete the physical activity bout and then remain in a seated position until 2-hours has passed since ingesting the meal. After this time they may leave the lab. Resting and post-activity heart rate and blood pressure will be recorded.

After the final trial, the accelerometer and continuous glucose monitoring devices will be collected and the participant's role in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Body Mass Index 18-30 kg/m2.
* Generally healthy.

Exclusion Criteria:

* Smoking.
* Pregnancy, or planning to become pregnant, or a nursing mother.
* More than 2 kg weight change during the last month.
* Diabetes.
* Evidence of, or being treated for, cancer or infectious/non-infectious chronic hematological, pulmonary, cardiac, hepatic, renal, or gastrointestinal diseases.
* Any contraindication to exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose concentrations. | In all trials, postprandial blood glucose concentrations will be measured - the change from baseline (immediately prior to meal ingestion) 2-hours after meal ingestion.
  Continuous glucose monitoring (CGM; Dexcom G5 Mobile) will be used to measure the change in glucose levels from baseline.

SECONDARY OUTCOMES:
Postprandial blood glucose control (mean). | In all trials, postprandial glucose control will be measured between baseline (immediately prior to meal ingestion) and the end of the trial (2-hours after meal ingestion).
  Mean glucose levels will be derived from CGM-measurements.
Postprandial blood glucose control (standard deviation). | In all trials, postprandial glucose control will be measured between baseline (immediately prior to meal ingestion) and the end of the trial (2-hours after meal ingestion).
  The standard deviation of glucose levels will be derived from CGM-measurements.
Postprandial blood glucose control. | In all trials, postprandial glucose control will be measured between baseline (immediately prior to meal ingestion) and the end of the trial (2-hours after meal ingestion).
  The mean amplitude of glycemic excursions will be derived from CGM-measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, Edgbaston, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Solomon TPJ, Tarry E, Hudson CO, Fitt AI, Laye MJ. Immediate post-breakfast physical activity improves interstitial postprandial glycemia: a comparison of different activity-meal timings. Pflugers Arch. 2020 Feb;472(2):271-280. doi: 10.1007/s00424-019-02300-4. Epub 2019 Aug 8. PMID 31396757